CLINICAL TRIAL: NCT02895646
Title: Genomic Study of Genetic Polymorphisms Involved in Immediate Allergic Reactions to Beta-lactam Antibiotics
Acronym: PANGENOMIC-BL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/PHRC/PANGENOMIC/GUEANT/MS
Record Dates: First submitted 2016-09-05; First posted 2016-09-12 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-09

CONDITIONS: Beta-Lactams Allergy; Hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Beta-lactam antibiotic allergy: Diagnosis based on clinical symptomatology and skin test positive for allergen and negative for other drugs and substances. Skin tests are performed 6 weeks after allergic reaction.
  Interventions: Other: Collection of blood sample
- Control: No specific clinical investigation for control subjects
  Interventions: Other: Collection of blood sample

INTERVENTIONS:
Other: Collection of blood sample

SUMMARY:
Beta-lactam antibiotics include penicillin and cephalosporins and are among the most prescribed antibiotics. This category of drugs is the most involved in immediate allergic manifestations with 2% reactions in treated subjects and a fatal outcome in 1/50000 treatments. Reactions are IgE-mediated and have a considerable but unknown genetic origin, revealed by studies in groups of different ethnical origins in the same geographical region. There are also some families with a high frequency of allergic reactions without identified Mendelian inheritance.

The purpose of this study is to identify predictive risk factors associated to immediate allergic reactions against beta-lactam antibiotics with a pangenomic approach.

A secondary purpose is to identify rare predictive factors with homozygosity mapping and exome sequencing in various families with high risk of allergy to beta-lactam antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Allergy group: Immediate allergic reaction (less than 2 hours after drug administration) to an antibiotic of penicillin or cephalosporin groups
* Allergy group: Positive skin test (intradermal test) with a non-irritant dilution of antibiotic of penicillin or cephalosporin groups

Exclusion Criteria:

* Refusal of participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population having an immediate IgE-mediated hypersensibility to beta-lactam antibiotics and matched control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 2356 (Actual)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Analysis of genetic polymorphisms predictive of risk of beta-lactam immediate allergy | day 0
  Common (>10%) or rare (1-10%) genetic polymorphisms in patients with beta-lactam immediate allergy

SECONDARY OUTCOMES:
Analysis of allelic homozygosity linked to allergen response, in more than 2 allergic individuals of the same family | day 0
  Allelic homozygosity in one or more regions of genome with one or more genes involved in allergen response, in more than 2 individuals affected by beta-lactam allergy in the same family
Severity of allergic reaction | day 0
  evaluated during clinical examination
Reactivity to skin test | day 0
Serum concentration of specific IgE | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis GUEANT, Principal Investigator — Service de BBMNM, CHU Nancy / unité INSERM U954, Faculté de Médecine, 54500 Vandoeuvre Les Nancy

IPD SHARING:
Plan to Share IPD: No